CLINICAL TRIAL: NCT04254809
Title: Evaluating a Web-based Intervention for Reactions to Suicidal Thoughts
Brief Title: Evaluation of a Computerized Intervention for Learning to Re-Evaluate Suicidal Thoughts
Acronym: REST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Face-to-face appointments, which were required by the IRB for suicide risk evaluation, were suspended by the IRB during the COVID-19 pandemic. During this pause, the PI left the institution. Thus, all study activities were terminated.
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Joseph William Boffa, Principal Investigator, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019.28553
Record Dates: First submitted 2020-02-02; First posted 2020-02-05 (Actual); Results first posted 2021-12-03 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Suicidal Ideation
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: Participants are randomized upon enrollment to one of two conditions: Re-Evaluating Suicidal Thoughts (active condition) or Healthy Social Living (control condition).
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant are blind to condition randomization, as are clinicians who provide suicide risk assessments throughout the follow-up period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Re-Evaluating Suicidal Thoughts (Experimental): Participants in this condition will complete the experimental intervention at the baseline appointment.
  Interventions: Behavioral: Re-Evaluating Suicidal Thoughts
- Healthy Social Living (Sham Comparator): Participants in this condition will complete the sham control intervention at the baseline appointment, and given the option to complete the experimental intervention at the conclusion of the follow-up period.
  Interventions: Behavioral: Healthy Social Living

INTERVENTIONS:
Behavioral: Re-Evaluating Suicidal Thoughts — Re-Evaluating Suicidal Thoughts (REST) is a is a computerized intervention designed to mitigate the experiential avoidance of suicidal thoughts. Over the course of approximately 30 minutes, individuals are provided with psychoeducation regarding the incidence rate, origin, conceptualization, and misconceptions of suicidal thoughts. Empirical evidence is presented to provide a scientific understanding of suicidal thoughts, and is aided through the use of metaphors to make concepts more accessible to viewers. REST draws from therapeutic strategies rooted in cognitive behavioral therapy (CBT) and Acceptance and Commitment Therapy (ACT) to further suggest tips for accepting (cp. approving of) the occurrence of suicidal thoughts, and introduces mindfulness and acceptance strategies for coping with them.
  Arms: Re-Evaluating Suicidal Thoughts
Behavioral: Healthy Social Living — To control for potential effects of time and presentation of educational material on study outcome variables, participants randomized to the control intervention will complete a computerized psychoeducation program regarding the benefits of social support networks. Across approximately 20 minutes of audiovisual slides, participants are informed of the ways in which social connections buffer against loneliness and facilitate social learning, provided tips for expanding and maintaining their social network, and administered a brief quiz to assess for comprehension.
  Arms: Healthy Social Living

SUMMARY:
As rates of suicide have increased over the last several decades, research has identified that roughly two-thirds of individuals who attempt suicide do so within one year from the time that they begin to think about suicide. This suggests a greater need for interventions designed to specifically help individuals learn to cope with thoughts of suicide to interrupt the process by which thoughts may lead to suicidal behaviors (i.e, attempts).

This study aims to develop and test a novel intervention designed to help individuals feel more confident in their ability to manage thoughts of suicide. It is common that individuals with suicidal ideation may not understand where thoughts of suicide come from and are therefore distressed at the prospect they might never escape these thoughts. As a result, these individuals may attempt to distract from or avoid these thoughts in ways that contribute to suicidal ideation becoming more frequent and intense over the long-term. This 'experiential avoidance' of suicidal ideation is therefore an excellent target for treatment and has in fact been shown to help reduce the distress associated with suicidal thoughts in several treatment studies.

The intervention to be tested in this study seeks to reduce the distress related to suicidal thoughts by explaining that these thoughts are a normative response to extreme stress, and provides strategies that help individuals observe that suicidal thoughts are temporary (i.e., will not last "forever") and something they can tolerate without needing to rigidly control them. To maximize the potential of this intervention to help the largest number of individuals, it is entirely computerized and takes only 30 minutes to complete. This will help reduce many of the traditional barriers to treatment that individuals with suicidal ideation face (e.g., costs, time restrictions, and stigma of help-seeking).

Individuals (N=106) with current suicidal ideation will be randomly assigned to participate in either the experiential avoidance intervention for suicidal thoughts or a control intervention. Experiential avoidance (i.e., distress or avoidance) and severity of suicide risk will be measured one week, and one month after participants complete their assigned intervention. It is expected that, compared to controls, individuals who receive the experiential avoidance intervention will report: 1) less experiential avoidance at one week follow-up, and 2) less severe suicide risk at one-month follow-up.

DETAILED DESCRIPTION:
Each year in the United States nearly 47,000 people die by suicide. Despite over 50 years of suicide prevention research, the field is no closer to identifying specific factors which influence the transition of suicidal ideation to suicide attempts. Research suggests upwards of 60% of individuals with suicidal ideation progress to making suicide plans or attempts within 1 year, suggesting a specific, pernicious process is involved in this escalation. Identifying which mechanisms contribute to the escalation of new-onset suicidal ideation is crucial to developing interventions that target these underlying processes.

Conceptual models of suicide have long viewed suicidal ideation and behaviors as a form of escape or avoidance from psychological distress with which individuals do not know how to cope. Indeed, psychiatric disorders are roughly 4 times as prevalent among suicidal ideators compared to non-ideators, and it is estimated 90% of suicide decedents evinced at least one psychiatric disorder. Several empirical models of psychiatric disorders implicate behavioral or experiential (i.e., emotional) avoidance as a driving mechanism of symptom severity (i.e., psychological distress. Similar to other psychiatric symptoms, suicidal ideation is distressing insofar as some individuals view such thoughts as incompatible with their natural instinct for self-preservation. To the extent that individuals respond to suicidal ideation with avoidance, such responses may in part be responsible for the escalation of suicidal ideation to plans or attempts.

Incidentally, models of psychological flexibility indicate a primary role for experiential avoidance and have been applied to suicidal ideation and behaviors. Higher levels of experiential avoidance are prospectively and concurrently associated with suicidal thoughts and behaviors. Moreover, as a cognitive-behavioral indicator of experiential avoidance, efforts to avoid or suppress suicidal thoughts are associated with greater concurrent levels of suicidal ideation and risk, and relate to a paradoxical increase in the severity of suicidal ideation over time.

Taken together, these studies suggest that individuals high in experiential avoidance with concomitant suicidal ideation may benefit from interventions that mitigate experience avoidance. Such interventions would ideally limit the psychological distress associated with the occurrence of suicidal thoughts, and improve one's ability to adaptively cope with suicidal thoughts rather than seeking to avoid, control, or suppress such thoughts. Indeed, preliminary evidence suggests treatment modalities that incorporate this approach (i.e., Acceptance and Commitment Therapy [ACT]) reduce suicidal ideation. Unfortunately, as with most traditional psychotherapies, this evidence stems from studies that required participants to attend numerous in-person sessions with a trained psychotherapist. Outside of treatment studies, the time and costs associated with this treatment would likely serve as a barrier to individuals with suicidal ideation, who represent a segment of the population that critically underutilize these types of mental health services. In order to increase suicide prevention efforts, it would be beneficial to develop ACT-based interventions that are more scalable and thus have the potential to address the needs of a greater number of individuals with suicidal ideation.

The current study therefore aims to develop and test a brief, web-based intervention primarily focused on reducing experiential avoidance of suicidal ideation among individuals with current SI (N = 106). The study will consist of one baseline appointment (in person), and two follow-up appointments one week (phone/online) and one month (phone/online) following their baseline appointment. At the baseline appointment, participants will complete measures of suicidal ideation severity and experiential avoidance. They will then be randomized to complete either the computerized experiential avoidance intervention or a healthy living control video safety planning with a clinician. Per best practices for maintaining participant safety, following intervention condition, all participants will receive the Safety Planning Intervention. One week after the baseline appointment, participants will complete a suicide risk assessment over the telephone, during which time they will also complete self-report measures of experiential avoidance and suicidal ideation severity. These same procedures will be conducted again one month after baseline.

It is hypothesized that, compared to healthy living controls, individuals who receive the experiential avoidance intervention will report: 1) less experiential avoidance at one week follow-up, and 2) less severe suicidal ideation at one-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Suicidal ideation during the past two-weeks

Exclusion Criteria:

* Imminent risk for attempting suicide, requiring hospitalization
* Unmedicated psychotic spectrum or bipolar disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Boffa, MS, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Re-Evaluating Suicidal Thoughts | Healthy Social Living
Started | 48 | 48
Completed | 43 | 38
Not Completed | 5 | 10
Not completed — Lost to Follow-up | 5 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Re-Evaluating Suicidal Thoughts | Healthy Social Living | Total
Number analyzed (Participants) | 48 | 48 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.54 (2.53) | 19.29 (2.42) | 19.42 (2.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 39 | 77
  Male | 10 | 9 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 15 | 29
  Not Hispanic or Latino | 34 | 33 | 67
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 5 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 6 | 14
  White | 32 | 41 | 73
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 48 | 48 | 96
Patient Health Questionnaire-8 [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionnaire-8 (PHQ-8) is a sum-scored measure of eight items which reflect the past two-week severity of depression symptoms. Total scores range from 0-24. Greater scores mean greater depression symptom severity.
  units on a scale | 20.85 (5.50) | 22.54 (5.62) | 21.70 (5.59)

OUTCOME MEASURES:

1. Primary Outcome: Standardized Residual Change in Experiential Avoidance of Suicidal Ideation
Description: Data sourced from Acceptance and Action Questionnaire for Suicidal Ideation (AAQ-SI) self-report measure total scores. AAQ-SI scores range from 4-28, higher scores indicate greater experiential avoidance of suicidal ideation. Standardized residual change calculated by regressing AAQ-SI scores at one week onto AAQ-SI scores at baseline. Positive values mean experiential avoidance of suicidal ideation increased relative to rest of sample. Negative values mean it decreased relative to rest of sample. Values follow a normal distribution, with nearly all falling between -3 and +3.
Time Frame: Baseline and One week
Population: Intention to treat analyses carried last observation forward for all participants enrolled at baseline.
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Re-Evaluating Suicidal Thoughts | Healthy Social Living
Number analyzed (Participants) | 48 | 48
Unitless | -0.32 (0.88) | 0.32 (1.01)
Statistical Analysis 1: Comparison: Re-Evaluating Suicidal Thoughts vs Healthy Social Living; Intention to treat analyses carried last observation forward for all participants enrolled at baseline. Standardized residual change score calculated by regressing scores at one-week follow-up onto scores at baseline; Test type: Superiority; p = .001, Regression, Linear — Threshold for statistical significance was p = .05; Slope = -0.64, 95% CI 2-sided [-1.02 to -0.25], Standard Error of Mean 0.19 — REST coded as 0, HSL coded as 1; negative slope reflects greater standardized reductions in outcome among REST compared to HSL

2. Primary Outcome: Standardized Residual Change in Suicide Risk Severity
Description: Data sourced from Beck Scale for Suicidal Ideation (BSS) self-report measure total score. BSS scores range from 0-38, higher scores indicate greater suicide risk severity. Standardized residual change calculated by regressing BSS scores at one month onto BSS scores at baseline. Positive values mean suicide risk severity increased relative to rest of sample. Negative values mean it decreased relative to rest of sample.
Time Frame: Baseline and one month
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Re-Evaluating Suicidal Thoughts | Healthy Social Living
Number analyzed (Participants) | 48 | 48
Unitless | -0.31 (0.87) | 0.31 (1.03)
Statistical Analysis 1: Comparison: Re-Evaluating Suicidal Thoughts vs Healthy Social Living; Intention to treat analyses carried last observation forward for all participants enrolled at baseline. Standardized residual change score calculated by regression scores at one-month follow-up onto scores at baseline; Test type: Superiority; p = .002, Regression, Linear — Threshold for significance was p = .05; Slope = -0.61, 95% CI 2-sided [-0.99 to -0.23], Standard Error of Mean 0.19 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Standardized Residual Change in Cognitive Avoidance of Suicidal Ideation
Description: Data sourced from White Bear Suppression Inventory for Suicidal Ideation (WBSI-SI) self-report measure distraction and suppression subscale score. WBSI-SI avoidance subscale scores range from 7-35, higher scores indicate greater cognitive avoidance of suicidal ideation. Standardized residual change calculated by regressing WBSI-SI avoidance scores at one week onto WBSI-SI avoidance scores at baseline. Positive values mean cognitive avoidance of suicidal ideation increased relative to rest of sample. Negative values mean it decreased relative to rest of sample.
Time Frame: Baseline and One week
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Re-Evaluating Suicidal Thoughts | Healthy Social Living
Number analyzed (Participants) | 48 | 48
Unitless | -.23 (1.18) | 0.23 (0.71)
Statistical Analysis 1: Comparison: Re-Evaluating Suicidal Thoughts vs Healthy Social Living; Intention to treat analyses carried last observation forward for all participants enrolled at baseline. Standardized residual change score calculated by regression scores at one-week follow-up onto scores at baseline; Test type: Superiority; p = .03, Regression, Linear — Threshold for statistical significance was p = .05; Slope = -0.45, 95% CI 2-sided [-0.86 to -.05], Standard Error of Mean .20 — REST coded as -, HSL coded as 1; negative slope reflects greater standardized reductions in outcome among REST compared to HSL

ADVERSE EVENTS:
Time Frame: Up to one month follow-up.
Arm/Group | Re-Evaluating Suicidal Thoughts | Healthy Social Living
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 0/48 | 0/48

LIMITATIONS AND CAVEATS:
Early termination prevented achieving recruitment target, but total number analyzed still exceeded the sample size necessary to detect medium effects in a priori power analysis. Intention-to-treat with lost observation carried forward was used to handle missing data and may not account for true scores at follow-up. However, the same pattern of results held for experiential avoidance and suicidal ideation severity among a completer sample. Those results are available upon request from the PI.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-27): https://cdn.clinicaltrials.gov/large-docs/09/NCT04254809/Prot_SAP_000.pdf